CLINICAL TRIAL: NCT03139578
Title: Short-Term Clinical Comparison of Two Silicone Hydrogel Daily Disposable Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR-5932
Record Dates: First submitted 2017-05-02; First posted 2017-05-04 (Actual); Results first posted 2018-12-11 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Visual Acuity

STUDY DESIGN:
Intervention Model Description: Contra-lateral Assignment
Who Masked: Participant, Investigator
Masking Description: Both the investigator and the subjects are masked to the identity of the study lenses. Lenses were over-labelled and coded to mask the lens foil. Over-labelling was carried out by the study sponsor following specific SOPs (see ICH GCP guidelines Section 5.13).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- C 8.5\C 9.0\T 8.5\T 9.0 (Experimental): Subjects randomized to this sequence received Control lens (base curve 8.5 on the left eye and 9.0 on the right eye) during the first period and then received Test lens (base curve 8.5 on the left eye and 9.0 on the right eye) during the second period.
  Interventions: Device: Test 8.5BC; Device: Test 9.0BC; Device: Control 8.5BC; Device: Control 9.0BC
- C 9.0\C 8.5\T 9.0\T 8.5 (Experimental): Subjects randomized to this sequence received Control lens (base curve 9.0 on the left eye and 8.5 on the right eye) during the first period and then received Test lens (base curve 9.0 on the left eye and 8.5 on the right eye) during the second period.
  Interventions: Device: Test 8.5BC; Device: Test 9.0BC; Device: Control 8.5BC; Device: Control 9.0BC
- T 8.5\T 9.0\C 8.5\C 9.0 (Experimental): Subjects randomized to this sequence received Test lens (base curve 8.5 on the left eye and 9.0 on the right eye) during the first period and then received Control lens (base curve 8.5 on the left eye and 9.0 on the right eye) during the second period.
  Interventions: Device: Test 8.5BC; Device: Test 9.0BC; Device: Control 8.5BC; Device: Control 9.0BC
- T 9.0\T 8.5\C 9.0\C 8.5 (Experimental): Subjects randomized to this sequence received Test lens (base curve 9.0 on the left eye and 8.5 on the right eye) during the first period and then received Control lens (base curve 9.0 on the left eye and 8.5 on the right eye) during the second period.
  Interventions: Device: Test 8.5BC; Device: Test 9.0BC; Device: Control 8.5BC; Device: Control 9.0BC

INTERVENTIONS:
Device: Test 8.5BC — senofilcon A contact lenses with 8.5 base curve
Device: Test 9.0BC — senofilcon A contact lenses with 9.0 base curve
Device: Control 8.5BC — narafilcon A contact lenses with 8.5 base curve
Device: Control 9.0BC — narafilcon A contact lenses with 9.0 base curve

SUMMARY:
This will be a 2 period one-day, double-masked, randomized, repeated measures, non-dispensing, cross-over study where the main purpose of this study is to compare the performance of a new daily disposable silicone hydrogel lens with that of an existing similar lens.

ELIGIBILITY:
Inclusion Criteria:

Potential subjects must satisfy all of the following criteria to be enrolled in the study:

1. The subject must read and sign the Informed Consent form.
2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. Healthy adult males or females aged 18-55 years.
4. The subject's spherical contact lens requirement in the range +2.00 D to +4.00 D or -1.00 D to -6.00 D.
5. The subject's refractive cylinder must be ≤1.00 D in each eye.
6. The subject must have visual acuity best correctable to 6/9 (20/30) or better for each eye.
7. The subject is a current soft contact lens wearer (defined as a minimum of 6 hours of DW per day, at least 5 days per week, for a minimum of 1 month prior to the study).
8. The subject must have normal eyes (i.e., no ocular medications or infections of any type).

Exclusion Criteria:

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

1. Currently pregnant or lactating
2. Any systemic disease (e.g., Sjögren's Syndrome),allergies, infectious disease (e.g., hepatitis,tuberculosis), contagious immunosuppressive diseases (e.g., HIV), autoimmune disease (e.g. rheumatoid arthritis), or other diseases, by self-report, which are known to interfere with contact lens wear and/or participation in the study.
3. Use of systemic medications (e.g., chronic steroid use) that are known to interfere with contact lens wear.
4. Any ocular allergies, infections or other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but not be limited to entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or corneal distortion.
5. Extended wear contact lens correction.
6. Any current use of ocular medication.
7. Any previous, or planned (during the course of the study) ocular surgery (e.g., radial keratotomy, PRK, LASIK, etc.)
8. Any greater than Grade 2 slit lamp findings (e.g., oedema, corneal neovascularisation, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA classification scale or any other ocular abnormality that may contraindicate contact lens wear.
9. Any contact lens-related history or signs of a corneal inflammatory event, or any other ocular abnormality that would contraindicate contact lens wear.
10. Participation in any contact lens or lens care product clinical trial within 14 days prior to study enrolment.
11. Employee, relative or friends of employees of any ophthalmic company, or investigational clinic (e.g., Investigator, Coordinator, Technician).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2017-04-28 (Actual); Primary Completion 2017-10-22 (Actual); Study Completion 2017-10-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Aston University Optometry and Vision Science, Birmingham
  - Visioncare Research, Farnham

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 51 subjects were enrolled in the study from two sites. Of those enrolled, 50 subjects were randomized and 50 subjects were dispensed a study lens. All 50 subjects completed the study, while no one discontinued from the study.
Period: Period 1
Arm/Group | C 8.5\C 9.0\T 8.5\T 9.0 | C 9.0\C 8.5\T 9.0\T 8.5 | T 8.5\T 9.0\C 8.5\C 9.0 | T 9.0\T 8.5\C 9.0\C 8.5
Started | 12 | 13 | 12 | 13
Discontinued | 0 | 0 | 0 | 0
Completed | 12 | 13 | 12 | 13
Not Completed | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | C 8.5\C 9.0\T 8.5\T 9.0 | C 9.0\C 8.5\T 9.0\T 8.5 | T 8.5\T 9.0\C 8.5\C 9.0 | T 9.0\T 8.5\C 9.0\C 8.5
Started | 12 | 13 | 12 | 13
Discontinued | 0 | 0 | 0 | 0
Completed | 12 | 13 | 12 | 13
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: All subjects who were administered any test article excluding subjects who drop out prior to administering any test article
Arm/Group | Total
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.3 (13.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 47
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 14
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 20
  More than one race | 13
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: Participants]
  United Kingdom | 50

OUTCOME MEASURES:

1. Primary Outcome: Overall Fit Acceptance
Description: Overall lens fit acceptance was assessed by the investigator based on lens fitting characteristics and graded on a scale of 0 to 5, where 0=should not be worn and 5=perfect fit. The score ranges from 0 to 5, where higher scores indicate better fitting. The number of eye for each Grade was reported.
Time Frame: 30-45 minutes after lens settling
Population: All subjects who had successfully completed all required assessments visits without any a major protocol deviations.
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Groups:
- Test 8.5BC: Subjects randomized to receive senofilcon A lens 8.5 base curve in either the right or left eye and successfully completed all assessments without a major protocol deviation.
- Test 9.0BC: Subjects randomized to receive senofilcon A lens 9.0 base curve in either the right or left eye and successfully completed all assessments without a major protocol deviation.
- Control 8.5BC: Subjects randomized to receive narafilcon A lens 8.5 base curve in either the right or left eye and successfully completed all assessments without a major protocol deviation.
- Control 9.0BC: Subjects randomized to receive narafilcon A lens 9.0 base curve in either the right or left eye and successfully completed all assessments without a major protocol deviation.
Arm/Group | Test 8.5BC | Test 9.0BC | Control 8.5BC | Control 9.0BC
Number analyzed (Participants) | 48 | 48 | 48 | 48
Number analyzed (Eyes) | 48 | 48 | 48 | 48
Eyes
  0 | 0 | 0 | 0 | 0
  1 | 0 | 0 | 0 | 0
  2 | 1 | 2 | 1 | 5
  3 | 5 | 8 | 5 | 7
  4 | 17 | 24 | 19 | 17
  5 | 25 | 14 | 23 | 19
Statistical Analysis 1: Comparison: Test 8.5BC vs Control 8.5BC; Test type: Non-Inferiority — Non-inferiority margin of 0.625 was used. If the lower limit of 95% confidence interval was greater than a non-inferiority margin of 0.625, then non-inferiority of Test relative to Control was concluded; Generalized linear mixed model; Simulation-based adjustment was utilized to address the multiple comparisons of different base curves; Cumulative Odds Ratio = 1.18, 95% CI 2-sided [0.46 to 3.06] — Cumulative odds ratio was calculated as Test over Control
Statistical Analysis 2: Comparison: Test 9.0BC vs Control 9.0BC; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Generalized linear mixed model; Simulation-based adjustment was utilized to address the multiple comparisons of different base curves; Cumulative Odds Ratio = 0.93, 95% CI 2-sided [0.34 to 2.52] — Cumulative odds ratio was calculated as Test over Control

2. Primary Outcome: Lens Power Requirement
Description: The lens power requirements (aka sphere requirements) for each lens type was calculated by summing the lens power and the spherical over-refraction. Then the difference of lens power requirement between the Test and Control lenses was calculated (Test-Control).
Time Frame: 30-45 minutes after lens settling
Population: All subjects who had successfully completed all required assessments without a major protocol deviation.
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Test 8.5BC | Test 9.0BC | Control 8.5BC | Control 9.0BC
Number analyzed (Participants) | 48 | 48 | 48 | 48
Number analyzed (Eyes) | 48 | 48 | 48 | 48
Eyes
  <= -3.75 | 10 | 9 | 10 | 8
  -3.50 to -3.00 | 7 | 9 | 7 | 10
  -2.75 to -2.25 | 17 | 15 | 16 | 15
  -2.00 t -1.50 | 9 | 10 | 10 | 10
  -1.25 to -0.75 | 2 | 2 | 3 | 2
  >= -0.50 | 3 | 3 | 2 | 3
Statistical Analysis 1: Comparison: Test 9.0BC vs Control 9.0BC; Test type: Equivalence — Equivalence margin of 70% was used for no difference in lens power requirement; Wilson Method; Proportion (%) = 93.8, 97.5% CI 2-sided [81.1 to 98.1] — Lens power requirement difference was calculated as Test minus Control. Then the proportion of eyes with similar lens power requirements (no difference or difference within ±0.25D) was calculated
Statistical Analysis 2: Comparison: Test 8.5BC vs Control 8.5BC; Test type: Equivalence — Equivalence margin of 70% was used for no difference in lens power requirement; Wilson Method; Proportion (%) = 83.3, 97.5% CI 2-sided [68.3 to 92.1] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Test 9.0BC vs Control 9.0BC; Test type: Equivalence — Equivalence margin of 80% was used for the lens power requirement difference within ±0.25 D; Wilson Method; Proportion (%) = 100, 97.5% CI 2-sided [90.5 to 100] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Test 8.5BC vs Control 8.5BC; Test type: Equivalence — Equivalence margin of 80% was used for the lens power requirement difference within ±0.25 D; Wilson Method; Proportion (%) = 100.0, 97.5% CI 2-sided [90.5 to 100.0] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Subjective Comfort at Lens Insertion
Description: Subjective comfort on insertion was assessed by the subject on an 11-point scale (0 to 10) where 0=painful and 10=can't be felt. The score ranges from 0 to 10, where higher scores indicate better comfort. The average comfort score for each lens was reported.
Time Frame: Immediately upon lens insertion
Population: All subjects who had successfully completed all required assessments without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Graded Scale 0-10
Units Other Than Participants: Eyes
Arm/Group | Test 8.5BC | Test 9.0BC | Control 8.5BC | Control 9.0BC
Number analyzed (Participants) | 48 | 48 | 48 | 48
Number analyzed (Eyes) | 48 | 48 | 48 | 48
Graded Scale 0-10 | 9.15 (1.353) | 9.04 (1.220) | 8.92 (1.302) | 9.02 (1.176)
Statistical Analysis 1: Comparison: Test 8.5BC vs Control 8.5BC; Test type: Non-Inferiority — Non-inferiority margin of -1 was used. If the lower limit of 95% confidence interval was greater than a non-inferiority margin of -1, then non-inferiority of Test relative to Control was concluded; Linear mixed model; Simulation-based adjustment was used to address the multiple comparisons; Least square mean difference = 0.2, 95% CI 2-sided [-0.3 to 0.7]
Statistical Analysis 2: Comparison: Test 9.0BC vs Control 9.0BC; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; Linear mixed model; Simulation-based adjustment was used to address the multiple comparisons; Least square mean difference = 0.0, 95% CI 2-sided [-0.5 to 0.5]

4. Secondary Outcome: Subjective Comfort After Lens Settling
Description: Subjective comfort on setting was assessed by the subject on an 11-point scale (0 to 10) where 0=painful and 10=can't be felt. The score ranges from 0 to 10, where higher scores indicate better comfort. The average comfort score for each lens was reported.
Time Frame: 30-45 minutes after lens settling
Population: All subjects who had successfully completed all required assessments without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Graded scale 0-10
Units Other Than Participants: Eyes
Arm/Group | Test 8.5BC | Test 9.0BC | Control 8.5BC | Control 9.0BC
Number analyzed (Participants) | 48 | 48 | 48 | 48
Number analyzed (Eyes) | 48 | 48 | 48 | 48
Graded scale 0-10 | 9.50 (0.715) | 9.27 (1.005) | 9.56 (0.769) | 9.13 (1.214)
Statistical Analysis 1: Comparison: Test 8.5BC vs Control 8.5BC; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; Linear mixed model; Simulation-based adjustment was used to address the multiple comparisons; Least square mean difference = -0.1, 95% CI 2-sided [-0.4 to 0.3]
Statistical Analysis 2: Comparison: Test 9.0BC vs Control 9.0BC; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; Linear mixed model; Simulation-based adjustment was used to address the multiple comparisons; Least square mean difference = 0.1, 95% CI 2-sided [-0.2 to 0.5]

5. Secondary Outcome: Subjective Vision Quality
Description: Subjective vision quality was assessed by the subject on an 11-point scale (0 to 10) where 0=extremely blurred and 10=perfect. The score ranges from 0 to 10, where higher scores indicate better vision quality. The average vision quality score for each lens was reported.
Time Frame: 30-45 minutes after lens settling
Population: All subjects who had successfully completed all required assessments without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Graded scale 0-10
Units Other Than Participants: Eyes
Arm/Group | Test 8.5BC | Test 9.0BC | Control 8.5BC | Control 9.0BC
Number analyzed (Participants) | 48 | 48 | 48 | 48
Number analyzed (Eyes) | 48 | 48 | 48 | 48
Graded scale 0-10 | 9.33 (0.753) | 9.25 (0.911) | 9.19 (1.104) | 9.19 (1.065)
Statistical Analysis 1: Comparison: Test 8.5BC vs Control 8.5BC; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; Linear mixed model; Simulation-based adjustment was used to address the multiple comparisons; Least square mean difference = 0.1, 95% CI 2-sided [-0.1 to 0.4]
Statistical Analysis 2: Comparison: Test 9.0BC vs Control 9.0BC; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; Linear mixed model; Simulation-based adjustment was used to address the multiple comparisons; Least square mean difference = 0.1, 95% CI 2-sided [-0.2 to 0.3]

6. Secondary Outcome: Subjective Handling
Description: Subjective handling was assessed by the subject on an 11-point scale (0 to 10) where 0=extremely difficult and 10=very easy. The score ranges from 0 to 10, where higher scores indicate better handling. The average handling score for each lens was reported.
Time Frame: Immediately upon lens insertion
Population: All subjects who had successfully completed all required assessments without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Graded scale 0-10
Units Other Than Participants: Eyes
Arm/Group | Test 8.5BC | Test 9.0BC | Control 8.5BC | Control 9.0BC
Number analyzed (Participants) | 48 | 48 | 48 | 48
Number analyzed (Eyes) | 48 | 48 | 48 | 48
Graded scale 0-10 | 9.17 (1.243) | 9.10 (1.242) | 9.13 (1.248) | 9.25 (1.139)
Statistical Analysis 1: Comparison: Test 8.5BC vs Control 8.5BC; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; Linear mixed model; Simulation-based adjustment was used to address the multiple comparisons; Least square mean difference = 0.0, 95% CI 2-sided [-0.5 to 0.5]
Statistical Analysis 2: Comparison: Test 9.0BC vs Control 9.0BC; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; Linear mixed model; Simulation-based adjustment was used to address the multiple comparisons; Least square mean difference = -0.1, 95% CI 2-sided [-0.6 to 0.4]

7. Secondary Outcome: Monocular High Contrast Visual Acuity (VA)
Description: Monocular high contrast distance VA with the study lenses was collected to the nearest letter using computer generated logMAR charts. 0.02 logMAR is equivalent to 1 letter. Negative logMAR values indicate better lens performance. The average visual acuity was reported for each lens type.
Time Frame: 30-45 minutes after lens settling
Population: All subjects who had successfully completed all required assessments without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | Test 8.5BC | Test 9.0BC | Control 8.5BC | Control 9.0BC
Number analyzed (Participants) | 48 | 48 | 48 | 48
Number analyzed (Eyes) | 48 | 48 | 48 | 48
logMAR | -0.02 (0.068) | -0.02 (0.083) | -0.02 (0.064) | -0.02 (0.061)
Statistical Analysis 1: Comparison: Test 8.5BC vs Control 8.5BC; Test type: Non-Inferiority — Non-inferiority margin of 0.1 was used. If the upper limit of 95% confidence interval was lower than a non-inferiority margin of 0.1, then non-inferiority of Test relative to Control was concluded; Linear mixed model; Simulation-based adjustment was used to address the multiple comparisons; Least square mean difference = 0.002, 95% CI 2-sided [-0.009 to 0.012]
Statistical Analysis 2: Comparison: Test 9.0BC vs Control 9.0BC; Test type: Non-Inferiority — [test comment as in outcome 7, analysis 1]; Linear mixed model; Simulation-based adjustment was used to address the multiple comparisons; Least square mean difference = -0.001, 95% CI 2-sided [-0.012 to 0.009]

ADVERSE EVENTS:
Time Frame: Throughout the entire duration of the study, approximately 1 day per subject.
Arm/Group | Test 8.5BC | Test 9.0BC | Control 8.5BC | Control 9.0BC
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50 | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-14): https://cdn.clinicaltrials.gov/large-docs/78/NCT03139578/Prot_SAP_000.pdf